CLINICAL TRIAL: NCT04752982
Title: A Feasibility Study of a Computerised Spatial Inattention Grasping Home-based Therapy for Stroke Survivors (c-SIGHT)
Brief Title: Can we Use c-SIGHT for Spatial Neglect in Stroke Survivors' Homes?
Acronym: c-SIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: Norwich Clinical Trials Unit, UK (Unknown); The Stroke Association, United Kingdom (Other)
Responsible Party: Principal Investigator, Stephanie Rossit, Lecturer, University of East Anglia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R207146; SA PGF 19/100016 (Other Grant/Funding Number: Stroke Association)
Record Dates: First submitted 2021-02-07; First posted 2021-02-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Stroke; Spatial Neglect; Inattention
Keywords: Stroke; Spatial Neglect; c-SIGHT; Feasibility Trial; Telerehabilition; Home-based therapy; Attention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated (using minimisation) to either the active intervention or attentional control group. Minimisation will use the following parameters: age, days since stroke, side of hemisphere damaged, and neglect severity (measured using the star cancellation test).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The outcome assessor, stroke survivor, carer, research team and clinical care staff (e.g. GP) will be blinded to group allocation. Participants will not be told if they are in the active or attentional control c-SIGHT group. The set-up and equipment is the same between the two arms and only the instructions differ.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- c-SIGHT intervention (Active Comparator): Grasp, lift and balance three wooden rods of different lengths.
  Interventions: Behavioral: c-SIGHT intervention
- c-SIGHT attentional control (Sham Comparator): Grasp and lift three wooden rods of different lengths from one end only (no attempt to balance rods).
  Interventions: Behavioral: c-SIGHT attentional control

INTERVENTIONS:
Behavioral: c-SIGHT intervention — The c-SIGHT active intervention involves grasping, lifting and balancing wooden rods using the unaffected hand. C-SIGHT uses a training mat, three wooden rods of different lengths, a laptop (to run the computer program) and a small motion tracking sensor which records the user's session length and trials completed. The participant's existing television is used to present the program (connected to the laptop).
  Arms: c-SIGHT intervention
Behavioral: c-SIGHT attentional control — The c-SIGHT attentional control exercises involves grasping and lifting wooden rods from one end using the unaffected hand. Identical to the intervention group, the c-SIGHT attentional control version uses a training mat, three wooden rods of different lengths, a laptop (to run the computer program) and a small motion tracking sensor which records the user's session length and trials completed. The participant's existing television is used to present the program (connected to the laptop).
  Arms: c-SIGHT attentional control

SUMMARY:
Spatial neglect is a common post-stroke condition in which people may not be aware of anything on one side of the world (usually the same side they lost their movement). Currently, there is no effective treatment for spatial neglect. A therapy called SIGHT (Spatial Inattention Grasping Home-based Therapy) has shown early evidence of improving stroke survivors' spatial neglect (Rossit et al., 2019). SIGHT involves individuals picking-up and balance wooden rods with their less affected hand, independently, without the need for a therapist present at all times. Working with stroke survivors, carers and clinicians we have developed of a computerized version of SIGHT (c-SIGHT; Morse et al., in press). The present trial aims to: 1) investigate the feasibility of a blinded randomized controlled trial of c-SIGHT (active intervention) vs. an attentional control training version of c-SIGHT (sham intervention) in the homes of stroke survivors with spatial neglect; 2) Explore participant's experience using c-SIGHT independently at home; and 3) Explore the potential effects and effect size of c-SIGHT active intervention compared to the attentional control training to inform a future Phase II trial.

DETAILED DESCRIPTION:
This is a multi-centre, two-arm blinded feasibility clinical trial with an embedded qualitative study. Following baseline assessment, participants will be randomized (using minimization) to either: active vs. sham version of computerised Spatial Inattention Grasping Home-based Therapy (c-SIGHT). Randomization and group allocation will be managed and run by Norwich Clinical Trials Unit (independent from research team and outcome assessors). Participants, carers, outcome assessors, clinical care team and research team will be blinded to participant group allocation. Participants allocated to the active intervention c-SIGHT group will be required to lift and balance three wooden rods of different lengths. Those in the attentional control c-SIGHT group will use the same equipment, but will be required to lift the rods from one end only and not attempt to balance them (an attentional control). During the first training session a therapist (independent from the outcome assessors) will set-up the equipment and train the participant to self-administer the relevant version of c-SIGHT independently (i.e., without the presence of a therapist). Following this training session, participants will self-administer the training for 10 consecutive days (thirty-minute sessions 2 times a day - 'Training phase'). On the last day of the training (day 10) the therapist will return to participant's homes to complete a monitoring visit and collect equipment. To monitor adherence and therapy compliance the therapist will collect photos and videos of the first and last session of the training. A blinded assessor will collect outcome assessments at the end of the training phase (T1) and at one-month post-training (T2). The post-training (T1) data collection visit will also include one-to-one semi-structured interviews with stroke survivor participants and their carers (qualitative study).

ELIGIBILITY:
Stroke survivors meeting all of the following criteria (and none of the exclusion criteria) at screening will be eligible to take part:.

* 18 years and older
* At least one-week post-stroke
* Stroke confirmed using clinical neuroimaging (head CT or MRI)
* Medically stable (as confirmed by the stroke service medical team responsible for the individual's stroke care)
* Capacity to give informed consent (as confirmed by the stroke service medical team responsible for the individual's stroke care and/or PI)
* Able to follow and execute a two-step command (e.g. "lift and balance this pen/pencil")
* Live within 70 miles of the University of East Anglia
* Signs of spatial neglect either via clinical assessment (e.g. star cancellation test; BIT) or observation

Exclusion criteria:

* History of other neurological conditions (e.g. dementia, brain tumour, Parkinson's disease, previous strokes)
* Bilateral impairment in arms (unable to move both arms)
* Taking part in a stroke rehabilitation research trial (which includes an intervention)

Carers must meet all the inclusion criteria to take part:

* 18 years and older
* Capacity to give informed consent
* Carer of stroke survivor in trial
* Live within 70 miles of the University of East Anglia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, approximately 2 years
  Rate of participants recruited into the trial amongst all participants screened
Exclusion rate | Through study completion, approximately 2 years
  Rate of participants excluded from participating amongst all participants screened
Attrition rate | Through study completion, approximately 2 years
  Rate of participants and data lost
Follow-up rate | Through study completion, approximately 2 years
  Rate of participants included at follow-up
Time required to collect and analyze data | Through study completion, approximately 2 years
  Time required for data collection and analysis will be computed per participant.
c-SIGHT compliance | 10 days
  Measured using short videos of participants carrying out first and final session of c-SIGHT. Following the participant's completion of the trial, videos will be reviewed by the research team to monitor whether participants and therapists deviated from instructions. Photo of set-up of first and last day of the training phase will also be checked to confirm set-up of equipment was correct and constant throughout the training phase.
Blinding and allocation success | Through study completion, approximately 2 years
  Evaluated by the frequency of unblinding occurred among stroke survivors, carers and outcome assessors and clinical care team. Success of allocation method using minimisation will be evaluated by measuring homogeneity of the two groups on co-variates such as age, time since stroke, hemisphere damage and neglect severity.
Adherence to c-SIGHT protocol | Through study completion, approximately 2 years
  The number of trials performed and length will be computed per session via a motion-tracking sensor.

SECONDARY OUTCOMES:
Star cancellation test | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  The Star Cancellation Test is a paper and pencil test developed to detect the presence of unilateral spatial neglect (USN) in the near extra personal space in patients with stroke.The maximum score that can be achieved on the test is 54 points. A cutoff of < 51 indicates the presence of SN. A Laterality Index or Star Ratio will be calculated from the ratio of stars cancelled on the contralesional side of the page and the total number of stars cancelled. Scores between 0 and 0.46 indicate neglect in the left hemispace. Scores between 0.54 and 1 indicate neglect in the right hemispace.This will be completed by stroke survivors only.
Line bisection test | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  A paper and pencil task that measures spatial biases when marking middle horizontal lines (10 lines of 20 mm length). The deviation in mm from center (bisection error) is averaged and a bisection error > that 6 mm is considered evidence of spatial inattention. Completed by stroke survivors only.
Computerised Extrapersonal Neglect Test (CENT) | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  Computerised visual search cancellation test and a line bisection test that measure spatial neglect in extra personal space via television screens. Stimuli are presented out of reach (e.g., on participant's television), run on a laptop and performed using a wireless remote. A variety of variables are produced including: total cancelled targets, allocentric and egocentric neglect scores, number of intersections and re-cancellations, quality of search, total time, time asymmetry, asymmetry accuracy, asymmetry search speed and bisection error. Formulas adapted from Dalmaijer et al. (2015). This outcome is completed by stroke survivors only.
  Completed by stroke survivors only.
Oxford Cognitive Screen | Baseline (T0, before intervention)
  The Oxford Cognitive Screen is a short cognitive screening tool specifically designed for stroke survivors inclusive for patients with aphasia and neglect. OCS returns scores and a visual snapshot of a patient's cognitive profile, in a 'wheel of cognition', which at a glance demonstrates the specific cognitive domain impairments in Attention, Language, Praxis, Number and Memory. Completed by stroke survivors only.
Broken Hearts test | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  Paper-and-pencil standardized measure of spatial neglect (part of Oxford Cognitive Screen). Number of targets and distractors cancelled as well as ego and allocentric scores will be computed. Completed by stroke survivors only.
Stroke Impact Scale (SIS) | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  The SIS is a stroke-specific, self-report, health status measure. It was designed to assess multidimensional stroke outcomes, including strength, hand function Activities of Daily Living / Instrumental Activities of Daily Living (ADL/IADL), mobility, communication, emotion, memory and thinking, and participation. An extra question on stroke recovery asks that the client rate on a scale from 0 - 100 how much the client feels that he/she has recovered from his/her stroke. Each item is rated using a 5-point Likert scale. Scoring will be computed for each domain and total according to scoring database: http://www.kumc.edu/school-of-medicine/population-health/research-and-community-engagement/stroke-impact-scale/instructions.html. Completed by stroke survivors only.
Spatial neglect visual analogue scale | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  A self-rating 10-point scale in which the participant will be asked to mark on a vertical line their (or their loved ones) perceived severity of spatial neglect. Completed by the stroke survivor and carer (if available) separately.
One item extended test | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  Observational test of contralesional limb awareness/personal neglect. Participants asked to point with unimpaired arm to six different parts of their body (e.g., ear, shoulder, elbow, side, leg, hand) and receive one of the following scores for each body part: 0 (no movement), 1 (search without reaching), 2 (reaching with hesitation and search), 3 (immediate reaching), with a total score ranging from 0 to 18. Completed by stroke survivors only.
Hand laterality task | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  Computerized task assessing body representation by testing perception of right vs. left hand images. Reaction times (ms) and errors (e.g., percentage) in identifying hands will be computed. Completed by stroke survivors only.
Body drawing task | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  Paper-and-pencil task requiring drawing of a person and self. Analysis will involve looking at symmetry of drawing and size/presence of different limbs. Completed by stroke survivors only.
1:1 semi-structured interview | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  Completed with the stroke survivor and carer (if available) separately. The interview, lasting approximately 15 minutes, will be transcribed and a thematic analysis will explore the usability of c-SIGHT and provide qualitative data about the therapy.
Modified Caregiver Strain Index | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  Questionnaire measuring financial, psychological, social, personal, physical caregiver strain. Carers indicate their agreement to statements from a choice three responses: 'Yes, on a regular basis' (2 points), 'Yes, sometimes' (1 point) and 'No' (0 points). Responses are summed and a higher score indicates greater strain. Completed by carer only (if available).
Catherine Bergego Scale (CBS) carer version | Baseline (T0, before intervention), post-training (T1, after 10 days of intervention) and at follow-up (T2, after 1 month post-training)
  The Catherine Bergego Scale is a standardized checklist to detect presence and degree of unilateral neglect during everyday life situations. The CBS uses a 4-point rating scale to report the frequency (e.g., Never, occasionally, frequently, always) of each statement occurring (e.g., "Forgets to groom/shave the left/right part of this/her face"). Responses are summed and the maximum score of 30 a total score of 30 indicates severe neglect. Completed by carer only (if available).
Rates of clinical brain scans obtained | Through study completion, approximately 2 years
  Number of clinical scans obtained.
System Usability Scale | Post-training (T1, after 10 days of intervention)
  To assess usability of c-SIGHT. Participants are asked to score the following 10 items with one of five responses that range from Strongly Agree to Strongly disagree. The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking. Based on previous research, a SUS score above 68 would be considered above average and anything below 68 is below average. This scale will be completed by the stroke survivor and carer (if available) separately.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Rossit, Ph.D, Principal Investigator — University of East Anglia
Locations (4):
- United Kingdom (4):
  - Cambridge University Hospital, Cambridge
  - Cambridgeshire and Peterborough NHS Foundation Trust, Cambridge
  - Norfolk & Norwich University Hospital NHS Foundation Trust, Norwich
  - Norfolk Community Health and Care NHS Trust, Norwich

IPD SHARING:
Plan to Share IPD: Yes
The final anonymised data set will be shared with other researchers through an open repository.
Supporting Information: Study Protocol
Time Frame: Study protocol will be published before or soon after recruitment has begun. The final, anonymised data set will be shared on an open repository (e.g., Open Science Framework) after the study has ended.
URL: https://osf.io/x2jg9/

REFERENCES:
- [Background] Rossit S, Benwell CSY, Szymanek L, Learmonth G, McKernan-Ward L, Corrigan E, Muir K, Reeves I, Duncan G, Birschel P, Roberts M, Livingstone K, Jackson H, Castle P, Harvey M. Efficacy of home-based visuomotor feedback training in stroke patients with chronic hemispatial neglect. Neuropsychol Rehabil. 2019 Mar;29(2):251-272. doi: 10.1080/09602011.2016.1273119. Epub 2017 Jan 24. PMID 28116988
- [Background] Morse H, Biggart L, Pomeroy V, Rossit S. Exploring perspectives from stroke survivors, carers and clinicians on virtual reality as a precursor to using telerehabilitation for spatial neglect post-stroke. Neuropsychol Rehabil. 2022 Jun;32(5):707-731. doi: 10.1080/09602011.2020.1819827. Epub 2020 Sep 18. PMID 32942950
- See also: Neurolab page for the trial (news, etc) — https://www.stephanierossit.com/c-sight